CLINICAL TRIAL: NCT05538572
Title: A Phase 1 Open-Label, Multi-Center, Safety and Efficacy Study of PRT3645 in Participants With Select Advanced or Metastatic Solid Tumors
Brief Title: A Study of PRT3645 in Participants With Select Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prelude Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRT3645-01
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer; Glioblastoma; Head and Neck Squamous Cell Carcinoma; Malignant Mesothelioma; Non-small Cell Lung Cancers; Sarcoma; Endometrial Cancer
Keywords: Advanced Solid Tumors; Breast Cancer; CDK4/6; Cyclin-dependent Kinase 4; Cyclin-dependent Kinase 6; Glioblastoma; Head and Neck Squamous Cell Carcinoma; HNSCC; Malignant Mesothelioma; Metastatic Solid Tumors; Non-small Cell Lung Cancers; NSCLC; PRT3645; Sarcoma; Endometrial Cancer
MeSH Terms: conditions — Breast Neoplasms; Glioblastoma; Squamous Cell Carcinoma of Head and Neck; Mesothelioma, Malignant; Sarcoma; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PRT3645 (Experimental): PRT3645 capsules will be self-administered once daily, continuously, at the dose-level assigned
  Interventions: Drug: PRT3645

INTERVENTIONS:
Drug: PRT3645 — PRT3645 capsules will be self-administered once daily, continuously, at the dose-level assigned

SUMMARY:
This is a Phase 1 dose-escalation study of PRT3645, a Cyclin-dependent Kinase 4/6 (CDK4/6) inhibitor, in patients with advanced or metastatic solid tumors. The purpose of this study is to investigate the safety, tolerability, dose limiting toxicity, and to determine maximally tolerated dose and recommended phase 2 dose to be used in subsequent development of PRT3645.

DETAILED DESCRIPTION:
This is an open-label, multicenter, dose-escalation Phase 1 study of PRT3645, a CDK4/6 inhibitor, evaluating patients with selected advanced or metastatic solid tumors including breast cancer (BC), glioblastoma (GBM), non-small cell lung cancer (NSCLC), sarcomas, head and neck squamous cell carcinoma (HNSCC), malignant mesothelioma, and endometrial cancer. The study plan expects to evaluate approximately eight dose levels however additional dose levels may be explored. Taking into account pharmacokinetic and pharmacodynamic data from the preceding dose levels, the dose may be escalated until a dose limiting toxicity is identified. Up to 15 patients may be enrolled at a dose shown to be tolerated for confirmation of the MTD and/or RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced, recurrent, or metastatic solid tumor malignancy that have either progress or ineligible for standard of care therapy:

  1. HR+ and HER2- or HR+ and HER2+ breast cancer
  2. Recurrent GBM (IDH wild type) or CDKN2A/B homozygous deleted IDH-mutant astrocytoma
  3. KRAS-mutant or SMARCA4 loss NSCLC
  4. CDK pathway alternation in any of the following tumor types: malignant mesothelioma, HPV-negative HNSCC (including oral cavity, oropharynx, hypopharynx, and larynx), sarcoma, or NSCLC
  5. Estrogen receptor positive with TP53 wild type endometrial cancer
* Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures
* Must have measurable or non-measureable (but evaluable) disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 or Karnofsky Performance Status (KPS) ≥80% (KPS is for GBM only)
* Adequate organ function.
* Able to swallow and retain oral medication.
* Must provide either archival or fresh tumor tissue sample during screening.

Exclusion Criteria:

* Participants with advanced, symptomatic, extensive visceral disease.
* Active inflammatory bowel disease or chronic diarrhea, short bowel syndrome, any upper gastrointestinal surgery including gastric resection, known malabsorption syndrome, or other condition that may impair absorption of PRT3645.
* Treatment with strong inhibitors of CYP3A4.
* History of another malignancy within 3 years except for adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancies, or malignancies previously treated with curative intent and not on active therapy or expected to require treatment or recurrence during the study.
* Clinically significant or uncontrolled cardiac disease, uncontrolled electrolyte disorders, uncontrolled or symptomatic CNS metastases or leptomeningeal disease except for GBM.
* Endometrial cancer patients who had received prior treatment with a CDK 4/6 inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) of PRT3645 | Baseline through Day 28
  Dose limiting toxicity will be evaluated over the 28-day observation period
Safety and tolerability of PRT3645: AEs, CTCAE Assessments | Baseline through approximately 2 years
  Safety and tolerability will be evaluated by incidence of DLTs, laboratory measurements, severity of adverse events (AEs) according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
Maximally tolerated dose (MTD)/Recommended phase 2 dose (RP2D) of PRT3645 | Baseline through approximately 2 years
  The MTD/RP2D will be established for further investigation in participants with advanced solid tumors

SECONDARY OUTCOMES:
Efficacy of PRT3645: Tumor assessment and responses | Baseline through approximately 2 years
  Objective response rate (ORR), Progression-free survival (PFS), Disease control rate (DCR) and Duration of response (DOR) will use RECIST v1.1, mRECIST v1.1, and/or RANO as primary measure for tumor assessment and response.
Pharmacokinetic profile of PRT3645: Minimum and maximum observed plasma concentration | Baseline through approximately 2 years
  PRT3645 pharmacokinetics will be calculated including the minimum and maximum observed plasma concentration.
Pharmacodynamic effect of PRT3645: Target engagement | Baseline through approximately 2 years
  Pharmacodynamic effect of PRT3645 demonstrating target engagement by assessment of phosphorylation of Rb.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (12):
  - Smilow Cancer Hospital Phase 1 Unit, New Haven, Connecticut
  - AdventHealth Medical Group Oncology Research at Celebration, Celebration, Florida
  - Miami Cancer Institute, Miami, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Laura and Isaac Perlmutter Cancer Center/ NYU Langone Health, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - NEXT Virginia, Fairfax, Virginia
- National Cancer Centre Singapore, Singapore, Singapore